CLINICAL TRIAL: NCT02107846
Title: A Phase 2a, Open-Label, Sequential Dose Escalation Study to Evaluate the Safety and the Pharmacokinetics of Oral PRX-112 (Plant Recombinant Human Glucocerebrosidase) in Enzyme Replacement Therapy-Naïve Subjects With Gaucher Disease
Brief Title: An Open-Label, Dose Escalation Study to Evaluate the Safety and the Pharmacokinetics of Oral PRX-112
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Protalix (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-112-02a
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 50 Units (Experimental): PRX-112 50 Units daily for 5 days
  Interventions: Drug: PRX-112
- 100 Units (Experimental): PRX-112 100 Units daily for 5 days
  Interventions: Drug: PRX-112
- 200 Units (Experimental): PRX-112 200 Units daily for 5 days
  Interventions: Drug: PRX-112
- 400 Units (Experimental): PRX-112 400 Units daily for 5 days
  Interventions: Drug: PRX-112

INTERVENTIONS:
Drug: PRX-112
  Other Names: Carrot Cells Expressing Recombinant Human Glucocerebrosidase

SUMMARY:
This is an open-label, dose escalation study to evaluate the safety of oral PRX-112 and pharmacokinetics of GCD in subjects with Gaucher disease naive to enzyme replacement therapy. The dose levels of PRX-112 are 50 units, 100 units, 200 units and 400 units GCD. Subjects will receive once daily oral administrations of PRX-112 for 5 consecutive days at each dose level with a 2-day washout period between doses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 or older
* Historical diagnosis of Gaucher disease by low leukocyte GCD activity level
* Haemoglobin ≥ 10 g/dL
* Body mass index (BMI) of 18 kg/m2-30 kg/m2 inclusive
* Subject is able to provide written informed consent
* Female subjects of child bearing potential must not be pregnant or lactating with a negative urine pregnancy test result at the screening visit.
* Female subjects of child-bearing potential and male subjects with female partners of childbearing potential must use two methods of contraception at all times during the study, one of which must be a barrier method. Acceptable methods of contraception are oral contraceptives, barrier methods (male condom, female condom, diaphragm, cervical cap, spermicide or intrauterine device), surgical sterility (documented doctor's report of vasectomy, hysterectomy and/or bilateral oophorectomy) and/or postmenopausal status (defined as at least 1 year without menses as demonstrated by medical history or subject report).
* Negative laboratory tests for HIV, HBsAg and HCV at the screening visit
* Naïve to any previous ERT or have received the last ERT treatment 12 months before signing IC

Exclusion Criteria:

* Presence of a gastrointestinal (GI) disease affecting motility or absorption
* Subjects with any history of allergic response to biological drugs or other allergies deemed clinically significant by the Investigator
* Reported history of alcohol or drug abuse
* Subject has donated blood in the 3 months prior to screening or subject has received plasma derivatives in the 6 months prior to screening
* Use of any investigational drug or participation in another clinical trial in the 3 months prior to screening (subject report)
* Subjects who have previously received ERT with positive anti-human plant recombinant GCD (prGCD) antibodies
* Clinical evidence of any active significant disease that could potentially compromise the ability of the Investigator to evaluate or interpret the effects of the study treatment on safety assessment, thus increasing the risk to the subject to unacceptable levels
* Presence of any medical, emotional, behavioural or psychological condition that, in the judgement of the Investigator, would interfere the compliance requirements of the study
* Subject has used any medication (excluding acetaminophen or dyprione) within 7 days of screening, including laxatives, teas and food additives known to be used for the treatment of constipation or diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve | 24 hours
  Blood samples for GCD level every 2 hours for 24 hours
Adverse Events | 7 Days
  Reporting of adverse events collected daily

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No